CLINICAL TRIAL: NCT00756015
Title: Healing After Arthroscopic Rotator Cuff Repair: A Prospective, Randomized Trial of Early Range of Motion Versus Immobilization
Brief Title: Post-op Rehabilitation's Influence on Tendon Healing & Clinical Outcomes Following Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Jay D. Keener, Assistant Professor Orthopaedic Surgery, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRPO 07-0915
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff; post-operative immobilization protocol; post-operative early motion protocol; physical therapy; cuff repair integrity; ultrasound
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Physical Therapy Modalities; Early Ambulation; Immobilization; Suburethral Slings

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Motion (Active Comparator): Other: Early range of motion post-operative therapy protocol.Early range of motion group: Shoulder pendulum exercises will be allowed from the time of surgery. Immediate range of motion of the elbow, forearm, wrist and hand. At the first postoperative visit, PROM of the shoulder will be permitted under therapist direction. Patients will avoid IR and behind the back stretching. At 6 weeks, AAROM and AROM will be advanced as tolerated. Capsular stretching will be advanced until full range of motion is achieved. Strengthening activities of the rotator cuff, deltoid and scapular stabilizers will be permitted at 3 months post surgery.
  Interventions: Other: Early Motion Protocol
- Immobilization (Other): Immobilization following rotator cuff repair.
  Interventions: Other: Immobilization

INTERVENTIONS:
Other: Early Motion Protocol — Early range of motion group: Shoulder pendulum exercises will be allowed from the time of surgery. Immediate range of motion of the elbow, forearm, wrist and hand. At the first postoperative visit, PROM of the shoulder will be permitted under therapist direction. Patients will avoid IR and behind the back stretching. At 6 weeks, AAROM and AROM will be advanced as tolerated. Capsular stretching will be advanced until full range of motion is achieved. Strengthening activities of the rotator cuff, deltoid and scapular stabilizers will be permitted at 3 months post surgery.
  Other Names: physical therapy; early mobilization
  Arms: Early Motion
Other: Immobilization — Immobilization group: 6 weeks of sling shoulder immobilization. Immediate range of motion of the elbow, forearm, wrist and hand. At 6 weeks, PROM and stretching of the shoulder allowed under therapist direction. At 12 weeks, AAROM and AROM exercises will be initiated and capsular stretching advanced until full ROM achieved. Strengthening activities of the rotator cuff, deltoid and scapular stabilizers will be permitted at 4 months post surgery.
  Other Names: Sling; Delayed active range of motion
  Arms: Immobilization

SUMMARY:
The purpose of this study is to better understand the influence of post-operative rehabilitation on the rate of tendon healing and clinical outcomes following arthroscopic repair of the rotator cuff. There are two schools of thought on what type of therapy program is most beneficial following surgical cuff repair. However there has been little data available to compare them. Therefore, the investigators would like to compare these two standard plans of care so that the investigators may better define the safety and efficacy of early mobilization of the shoulder versus keeping the shoulder immobilized following surgical management.

DETAILED DESCRIPTION:
Background

Rotator cuff disease is the leading cause of shoulder pain and disability. Previous studies regarding the epidemiology of rotator cuff disease have demonstrated a high incidence of age- related cuff tears, approximately 50% of individuals over the age of 55 years 1-3. Failure of conservative treatment often leads to surgical repair of the torn rotator cuff tendons. Indeed, rotator cuff repair is one of the most common surgical procedures currently performed in the shoulder with approximately 200,000 Americans undergoing this surgery yearly. We estimate that the Shoulder and Elbow Service at Washington University performs approximately 400 rotator cuff repairs per year.

One of the primary concerns following repair of the rotator cuff is healing of the repaired tendon. Although pain relief and improved shoulder function are predictable following rotator cuff repair, the rate of healing of the tendon repair has been much less consistent. In most instances, the repaired tissue is degenerative, 4, 5 possesses a poor blood supply 6 and, therefore, a limited ability to heal following repair. The rates of healing of the repaired cuff tendons have ranged from 6% to 80% across multiple studies depending on a variety of patient, tendon tear and surgery related factors 7-13. The major factors that have been identified to effect healing after rotator cuff repair include patient age, the size of the tear and the strength of the repair construct 8, 9, 12. To this point, there has been little data regarding the potential influence of postoperative rehabilitation of the shoulder on the structural integrity of rotator cuff repairs.

The Shoulder and Elbow Service at Washington University has had extensive experience in studying various factors related to not only the progression of rotator cuff disease, but also tendon healing and outcomes of treatment 8, 14-16. A strength of our research team has been the collaborative experience developed with musculoskeletal radiologists at the Mallinkrodt Institute using high-resolution ultrasound to examine the integrity of the rotator cuff. Extensive data with ultrasound at this institution has validated it as a highly accurate means of identifying and quantifying rotator cuff tears in both the preoperative and postoperative settings 17-20. High-resolution ultrasound, in the hands of experienced musculoskeletal radiologists, has been proven to be more accurate than magnetic resonance imaging in assessing the integrity of the rotator cuff in the postoperative setting 19. With this modality, we have been able to study the outcomes and tendon healing rates following repair of the rotator cuff using conventional arthroscopic repair techniques 8. Recent data, from this institution, has also been completed examining the clinical outcomes and repair integrity following newer arthroscopic techniques (double-row rotator cuff repairs) in three separate patient populations: partial thickness cuff tears, full thickness cuff tears and revision of recurrent rotator cuff tears (manuscripts in progress). Our service has also been currently involved in a NIH R01 funded study prospectively examining factors related to the progression of asymptomatic rotator cuff tears over time. Given our research experience with ultrasound, the Shoulder and Elbow Service at Washington University has been uniquely positioned to study one of the most important issues in shoulder surgery - the effect of rehabilitation on healing of the rotator cuff following surgical repair.

In addition to tendon healing, one of the primary goals following shoulder surgery is the early restoration of range of motion of the joint. Stiffness is one of the more common complications following shoulder surgery. Early range of motion helps to prevent the formation of adhesions within the joint and surrounding capsule and ligaments. Although most cuff repair constructs provide sufficient stability for early range of motion, the effect of motion at the repair site and the subsequent effect on healing are unknown in humans. Concerns regarding a deleterious effect of early motion on tendon healing have led some investigators to advocate substantially more conservative rehab after surgery. A delay in motion at the shoulder may theoretically improve the rate of tendon healing as stresses are minimized across the tendon repair site. This may be particularly important given that tendon repair constructs gradually becomes weaker before a more mature healing response occurs. However, a delay in motion will slow the return of mobility to the shoulder and may increase the risk of prolonged stiffness. Therefore, the clinician must balance the potential benefit (prevention of stiffness) against the potential harm (compromise of the surgical repair) of early rehabilitation following rotator cuff repair surgery. Despite the critical role early motion may have, there have been no published studies examining the influence of postoperative rehabilitation on the clinical outcomes and repair integrity following rotator cuff repair.

The primary purpose of this study is to examine the influence of postoperative rehabilitation on the rate of tendon healing and clinical outcomes following arthroscopic repair of the rotator cuff. The ideal rehabilitation protocols following rotator cuff repair have yet to be determined. The clinical impact of this study will be significant in that we will better define the safety and efficacy of early mobilization of the shoulder following the surgical management of rotator cuff tears. A better understanding of appropriate postoperative physical therapy regimens is fundamental to the effective care of patients following rotator cuff repair. This study will serve as a basis for further research defining nonsurgical factors that influence tendon healing and outcome after rotator cuff repair.

Specific Aim 1: To prospectively compare the rate of tendon healing following arthroscopic repair of small and medium sized tears of the rotator cuff in patients treated with two distinct postoperative rehabilitation protocols: immobilization versus early range of motion.

Hypothesis 1: The rate of tendon healing following repair of small to medium sized rotator cuff tears will be the same for those patients treated with immobilization compared to an early range of motion protocol.

Specific Aim 2: To prospectively compare the clinical outcomes following arthroscopic repair of small and medium sized tears of the rotator cuff in patients treated with two distinct postoperative rehabilitation protocols: immobilization versus early range of motion.

Hypothesis 2: The clinical results following repair of small to medium sized rotator cuff tears will be substantially better for those patients treated with an early range of motion protocol as compared to those that were immobilized.

A preliminary power analysis has been performed to determine the necessary number of patients for each group (alpha level =.05 and beta level = .20). Data from this institution suggests an 80% healing rate within this age group for small and medium size rotator cuff tears fixed with double-row cuff repair techniques. Given a presumed healing rate of 80% in the immobilization group, the numbers necessary to detect a difference in healing of 20% between the two rehabilitation protocols is 70 subjects in each group. Assuming a conservative attrition rate of 20%, we will estimate that a total of 170 subjects will need to be enrolled in this study.

All rotator cuff repairs will be performed with a standard technique utilizing arthroscopic double-row suture anchor constructs. The surgery will also include subacromial decompression and acromioplasty as dictated by acromial degenerative changes. Concomitant procedures related to the biceps tendon will be performed as indicated. At the time of preoperative surgical evaluation, patients will be randomized by sealed envelope into one of two postoperative rehabilitation groups:

Immobilization group: 6 weeks of sling shoulder immobilization. Immediate range of motion of the elbow, forearm, wrist and hand. At 6 weeks, PROM and stretching of the shoulder allowed under therapist direction. At 12 weeks, AAROM and AROM exercises will be initiated and capsular stretching advanced until full ROM achieved. Strengthening activities of the rotator cuff, deltoid and scapular stabilizers will be permitted at 4 months post surgery.

Early range of motion group: Shoulder pendulum exercises will be allowed from the time of surgery. Immediate range of motion of the elbow, forearm, wrist and hand. At the first postoperative visit, PROM of the shoulder will be permitted under therapist direction. Patients will avoid IR and behind the back stretching. At 6 weeks, AAROM and AROM will be advanced as tolerated. Capsular stretching will be advanced until full range of motion is achieved. Strengthening activities of the rotator cuff, deltoid and scapular stabilizers will be permitted at 3 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Full-thickness tears of the rotator cuff involving the supraspinatus that may or may not include the infraspinatus tendon (less than 25 mm anteroposterior dimension)
2. Arthroscopic double-row cuff repair

Exclusion Criteria:

1. Acute rotator cuff tears less than 6 weeks from injury
2. Subscapularis tendon tears (full thickness)
3. Preoperative stiffness: loss of greater than 30 passive elevation and/or ER compared to the opposite shoulder
4. Inability to comply with postoperative rehabilitation protocols
5. Inflammatory disease
6. Prior surgery of the shoulder

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of Shoulder function and strength | 3 months, 6 months, 1 year and 2 years post op

SECONDARY OUTCOMES:
Evaluation of cuff repair integrity using Ultrasound at 1 year post op | 1 year post op

CONTACTS AND LOCATIONS:
Overall Officials: Jay Keener, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine - Department of Orthopedics, St Louis, Missouri, United States